CLINICAL TRIAL: NCT02891720
Title: Feasibility of an Ingestible Sensor System to Measure PrEP Adherence in YMSM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hektoen Institute for Medical Research (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01AI122308 (NIH); R01AI122308 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A: Proteus Sensor System (PSS) First (Active Comparator): ARM A will receive Proteus Sensor System (PSS) first. At 12-week intervals participants will crossover to the next condition.
  Interventions: Device: Proteus Sensor System
- ARM B: SOC First (No Intervention): ARM B will 12 weeks of FTC/TDS standard of care (SOC) first. At 12-week intervals participants will crossover to the next condition.

INTERVENTIONS:
Device: Proteus Sensor System — The Proteus Sensor System (PSS) intervention includes 12 weeks of daily FTC/TDF with a weekly text messages transmitted to participants with estimated HIV risk reduction based upon the DBS algorithm.
  Arms: ARM A: Proteus Sensor System (PSS) First

SUMMARY:
The goal of this study is to evaluate an integrated technology system that confirms ingestion of oral PrEP, monitors adherence both in real-time and longitudinally, and provides visual feedback mechanisms to promote enhanced adherence behaviors.

DETAILED DESCRIPTION:
In order to evaluate the feasibility and acceptability of the PSS for FTC/TDF PrEP, 100 HIV-negative YMSM will be randomized in the Advances in Technology to Enhance Adherence Monitoring (A-TEAM) pilot study to 12 weeks of daily FTC/TDF with the PSS versus daily FTC/TDF standard-of-care (SOC), then each arm will crossover to 12 weeks of daily FTC/TDF without the sensor system versus with the sensor system, respectively. PrEP will be provided by the study (see Gilead letter) and other aspects of PrEP clinical care will be consistent with the PrEP Clinic's standard practices based on CDC clinical guidelines. The detection accuracy of the PSS will be correlated with DBS-determined TFV-DP and FTC-TP levels obtained monthly from participants. A relationship between TVF-DP in DBS and adherence to FTC/TDF PrEP in the preceding 1-3 months has previously been characterized. These adherence categories were implemented in iPrEx OLE and consisted of: below lower limit of quantitation (BLQ), >BLQ to 349 fmol per punch (fewer than two tablets per week), 350-699 fmol per punch (two or three tablets per week), 700-1249 fmol per punch (four to six tablets per week), and 1250 fmol per punch or more (daily dosing). Real-time visual feedback of medication ingestion will be provided to the participant via the PSS and transmitted to the study team. A weekly text message with estimated HIV risk reduction based upon the DBS algorithm will be transmitted to participants after the initial first week of FTC/TDF dosing. Finally, in-depth qualitative exploration of barriers and facilitators to use of the PSS components will be completed through individual interviews as well as focus group discussions with participants. Participants will also provide feedback on text messages regarding PrEP protection as well as suggestions for other potential methods to receive performance data.

ELIGIBILITY:
Inclusion Criteria

Young men who meet all of the following criteria are eligible for inclusion:

* PrEP-eligible YMSM
* Ages 18-24
* Biologically born male
* Report interest in PrEP
* Intend to use PrEP for a full 6 month period
* Eligible to be a PrEP patient at the CORE Center PrEP Clinic
* Meet one the following sexual risk criteria:

  * Have an HIV-positive sexual partner
  * Had recent bacterial STI
  * Report high numbers of sexual partners
  * Report history of inconsistent or no condom use
  * Report exchange/transactional sex.

Exclusion Criteria

Young men who meet any of the following criteria will be excluded:

* HIV+
* Creatinine clearance <60 cc/min)
* Allergy to topical adhesive
* Acute gastrointestinal symptoms
* History of major GI surgery
* Presence of an implanted electronic medical device.
* Subjects who are receiving any of the following medications:Nephrotoxic drugs (e.g., cidofovir, amphotericin, aminoglycosides, dapsone, tacrolimus, foscarnet, ACE inhibitors), all diuretics, drugs that may interfere with TFV excretion (e.g., (Val)ganciclovir, Cyclosporin A, Sirolimus, Antineoplastics), drugs (not including mineral and vitamin supplements) used for treatment of osteoporosis (e.g., alendronate and other bisphosphonates, teriparatide, denosumab, and calcitonin), chronic use of oral or systemic steroids (i.e., daily use for two weeks or more is not allowed), experimental medications that are not Food and Drug Administration (FDA)-approved, and FTC/TDF (Truvada®) received outside of the study

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of HIV-negative YMSM taking part in PSS intervention who adhere to PrEP medication | Up to 33 months

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will provide pharmacokinetic data along with evidence of the feasibility and acceptability of the novel Proteus adherence monitoring system for use among young MSM who are highly vulnerable to HIV infection. Audiences for dissemination are: 1) scientists; 2) primary and secondary prevention practitioners; and 3) YMSM, their partners, and their friends/families. Traditional dissemination vehicles will be used including manuscripts and presentations at international and national meetings. To facilitate integration of the findings into the public health arena, the protocol team will work closely with their YAB and present findings in forums attended by community-based organizations, such as local PrEP trainings and workshops.